CLINICAL TRIAL: NCT04353024
Title: Effects of Dimethyltryptamine (DMT) in Healthy Subjects: A Placebo-controlled Cross-over Study
Brief Title: Effects of Dimethyltryptamine in Healthy Subjects
Acronym: DMT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BASEC 2020-00376
Record Dates: First submitted 2020-04-06; First posted 2020-04-20 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Healthy
MeSH Terms: interventions — N,N-Dimethyltryptamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, 5-period cross-over design with 4 different doses of DMT and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Bolus of 0 mg DMT + perfusion of 0 mg/min DMT over 60 min, resulting in a total dose of 0 mg DMT.
  Interventions: Drug: Saline
- Low dose (Experimental): Intravenous bolus of 0 mg DMT + perfusion of 0.6 mg/min DMT over 90 min, resulting in a total dose of 54 mg DMT.
  Interventions: Drug: Dimethyltryptamine (DMT); Drug: Saline
- Low dose with bolus (Experimental): Intravenous bolus of 15 mg DMT + perfusion of 0.6 mg/min DMT over 90 min, resulting in a total dose of 69 mg DMT.
  Interventions: Drug: Dimethyltryptamine (DMT)
- High dose (Experimental): Intravenous bolus of 0 mg DMT + perfusion of 1 mg/min DMT over 90 min, resulting in a total dose of 90 mg DMT.
  Interventions: Drug: Dimethyltryptamine (DMT); Drug: Saline
- High dose with bolus (Experimental): Intravenous bolus of 25 mg DMT + perfusion of 1 mg/min DMT over 90 min, resulting in a total dose of 115 mg DMT.
  Interventions: Drug: Dimethyltryptamine (DMT)

INTERVENTIONS:
Drug: Dimethyltryptamine (DMT) — Intravenous DMT bolus and/or DMT maintenance perfusion over 90 min
  Arms: High dose; High dose with bolus; Low dose; Low dose with bolus
Drug: Saline — Intravenous saline bolus and/or saline maintenance perfusion over 90 min
  Arms: High dose; Low dose; Placebo

SUMMARY:
N,N-dimethyltryptamine (DMT) is a naturally-occurring psychedelic substance widely used in recreational and spiritual settings. DMT can be used as a tool to induce an altered state of consciousness of interest in psychological and psychiatric research. DMT is rapidly metabolized by monoamine oxidase (MAO) A. Therefore, it is inactive when administered orally and has a very short duration of action when administered parenterally (<20 min).Therefore, an intravenous administration regime including a bolus and maintenance perfusion has been proposed to induce a stable and prolonged DMT experience allowing to study the psychological and autonomic acute effects of DMT. This administration allows to induce and end an altered state safely and quickly. The goal of the present study is to experimentally test different intravenous DMT administration schedules to investigate the subjective and autonomic effects of DMT in healthy subjects.

DETAILED DESCRIPTION:
N,N-dimethyltryptamine (DMT) is a naturally-occurring psychedelic substance widely used in recreational and spiritual settings in the form of Ayahuasca. Similar to lysergic acid diethylamide (LSD) or psilocybin, DMT is considered a tool to induce an altered state of consciousness of interest in psychological and psychiatric research. Pharmacologically, DMT interacts with the serotonin 5-HT2A receptor similar to other classic hallucinogens including LSD and psilocybin. The main difference of DMT in comparison with LSD or psilocybin is inactivity when administered orally without monoamine oxidase (MAO) A inhibition and its short action when administered intravenously or by inhalation. In Ayahuasca, DMT is consumed iin combination with harmala alkaloids that inhibit MAO to increase the oral bioavailability of DMT and to prolong its action after oral use. Alternatively, an intravenous administration regime including a bolus and a one hour maintenance perfusion has been proposed to induce a stable and prolonged DMT experience, allowing to study the psychological and autonomic acute effects of DMT. Also, the maintenance perfusion administration allows to end an altered state of consciousness quickly. In the present study this model will be tested using four modified administration schemes. The goal of this study is to experimentally test different intravenous DMT administration schedules to investigate the subjective and autonomic effects of DMT in healthy subjects. The study is expected to inform researchers on dosing regimes of intravenous DMT as a tool to examine alterations of the mind and is of interest for psychology and psychiatry. This study does not intend to provide any therapeutic benefit for the participants. Currently, no study has validly determined the elimination half-life of DMT and other pharmacokinetic parameters. The key aim is to test the dose-response of DMT as well as the difference between the loading dose bolus and no-bolus perfusion conditions regarding pharmacokinetic, subjective, and autonomic effects including psychological and physical tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 65 years old
* Sufficient understanding of the German language
* Understanding of procedures and risks associated with the study
* Willing to adhere to the protocol and signing of the consent form
* Willing to refrain from the consumption of illicit psychoactive substances during the study
* Abstaining from xanthine-based liquids from the evenings prior to the study sessions and during the sessions
* Willing not to operate heavy machinery within 6 h of DMT administration
* Willing to use double-barrier birth control throughout study participation
* Body mass index between 18-29 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition
* Current or previous major psychiatric disorder
* Psychotic disorder or bipolar disorder in first-degree relatives
* Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
* Hallucinogenic substance use (not including cannabis) more than 20 times or any time within the previous two months
* Pregnancy or current breastfeeding
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medication that may interfere with the effects of the study medication
* Tobacco smoking (>10 cigarettes/day)
* Consumption of alcoholic beverages (>20 drinks/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Altered states of consciousness profile | 150 minutes
  Assessed once on each study day via 5 Dimensions of Altered States of Consciousness (5D-ASC) scale consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects
Subjective effect ratings over time | 150 minutes
  Assessed 22 times on each study day via Subjective Effect Scale (SES), consisting of 4 questions to be rated on a Likert scale ranging from 1 to 10, with higher ratings indicating stronger effects

SECONDARY OUTCOMES:
Subjective mood ratings | 150 minutes
  Assessed twice on each study day via the Adjective Mood Rating Scale (AMRS) consisting of 60 items to be rated on a 4-point Likert scale, with higher ratings indicating stronger identification with the specific mood
Mystical-type experiences | 150 minutes
  Assessed once on each study day via States of Consciousness Questionnaire (SCQ) which measures the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely")
Autonomic effects I | 150 minutes
  Assessed 22 times on each study day via systolic and diastolic blood pressure, Emax
Autonomic effects II | 150 minutes
  Assessed 22 times on each study day via heart rate, Emax
Plasma levels of DMT | 150 minutes
  Assessed 21 times on each study day via blood samples
Plasma levels of blood-derived neurotrophic factor (BDNF) | 150 minutes
  Assessed 21 times on each study day via blood samples
Plasma levels of oxytocin | 60 minutes
  Assessed twice on each study day via blood samples
Renal clearance of DMT | 3 hours
  Collected once per study day via one-time interval urine recovery
Effect moderation through personality traits I | Baseline
  Assessed via NEO-Five-Factor-Inventory (NEO-FFI)
Effect moderation through personality traits II | Baseline
  Assessed via Freiburger Personality Inventory (FPI)
Effect moderation through personality traits III | Baseline
  Assessed via Saarbrücker Personality Questionnaire (SPF)
Effect moderation through personality trait IV | Baseline
  Assessed via Elliot Humility Scale (EHS) which measures the personality trait humility through 13 items on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree"
Effect moderation through personality trait V | Baseline
  Assessed via Jankowski Humility Scale (JHS) which measures the personality trait humility through 18 items on a 5-point Likert scale ranging from "not at all" to "strongly"
Effect moderation through personality trait VI | Baseline
  Assessed via Arnett Inventory of Sensation Seeking (AISS-d)
Effect moderation through personality trait VII | Baseline
  Assessed via Defense Style Questionnaire (DSQ-40)
Adverse effects | 150 minutes
  Assessed via the List of Complaints (LC) which covers the emergence of 66 complaints in a yes/no format

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Basel-Stadt BS, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogt SB, Ley L, Erne L, Straumann I, Becker AM, Klaiber A, Holze F, Vandersmissen A, Mueller L, Duthaler U, Rudin D, Luethi D, Varghese N, Eckert A, Liechti ME. Acute effects of intravenous DMT in a randomized placebo-controlled study in healthy participants. Transl Psychiatry. 2023 May 23;13(1):172. doi: 10.1038/s41398-023-02477-4. PMID 37221177